CLINICAL TRIAL: NCT02459964
Title: A Randomized Trial to Compare Fentanyl Nasal Spray With Intravenous Opioids to Treat Severe Pain in Cancer Patients in the Emergency Department Setting
Brief Title: Compare Fentanyl Nasal Spray With Intravenous Opioids to Treat Severe Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-0086; NCI-2015-01509 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-05-29; First posted 2015-06-02 (Estimated); Results first posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Advanced Cancers; Pain
Keywords: Advanced Cancers; Pain; Fentanyl nasal spray; Hydromorphone hydrochloride; Phone call; Numeric Rating Scale; NRS
MeSH Terms: conditions — Pain | interventions — Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fentanyl Nasal Spray (Experimental): Fentanyl nasal spray 100 mcg delivered at time 0 (defined as the time when intranasal Fentanyl spray is administered) with a rescue dose allowed at time 0.5 hour (h).
  Study nurse to call patient 24 hours after participation to ask about side effects since taking part in the study.
  Interventions: Drug: Fentanyl Nasal Spray; Behavioral: Phone Call
- Hydromorphone Hydrochloride (Active Comparator): Hydromorphone hydrochloride 1.5 mg pushed intravenously (IV) at time 0 (defined as the time of completion of opioid IV push) with a rescue dose allowed at time 0.5 hour (h).
  Study nurse to call patient 24 hours after participation to ask about side effects since taking part in the study.
  Interventions: Drug: Hydromorphone Hydrochloride; Behavioral: Phone Call

INTERVENTIONS:
Drug: Fentanyl Nasal Spray — Fentanyl nasal spray 100 mcg delivered at time 0 (defined as the time when intranasal Fentanyl spray is administered) with a rescue dose allowed at time 0.5 hour (h)
  Arms: Fentanyl Nasal Spray
Drug: Hydromorphone Hydrochloride — Hydromorphone hydrochloride 1.5 mg pushed intravenously (IV) at time 0 (defined as the time of completion of opioid IV push) with a rescue dose allowed at time 0.5 hour (h).
  Arms: Hydromorphone Hydrochloride
Behavioral: Phone Call — Study nurse to call patient 24 hours after participation to ask about side effects since taking part in the study. The phone call should last about 5 minutes.

SUMMARY:
The goal of this clinical research study is to compare fentanyl nasal spray with a standard drug given by vein (hydromorphone hydrochloride) to help reduce pain related to cancer in patients coming to the emergency department.

DETAILED DESCRIPTION:
Study Groups and Drug Administration:

If participant agrees to take part in this study, they will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. This is done because no one knows if one study group is better, the same, or worse than the other group. Participant will have an equal chance of being in either group:

* If participant is in Group 1, they will receive the fentanyl nasal spray. The study staff will help participant use the nasal spray.
* If participant is in Group 2, the emergency center nurse will give them the hydromorphone hydrochloride by vein.

Study Procedures:

Participant will stay in the emergency department for at least 4 hours and will be monitored after receiving fentanyl or hydromorphone hydrochloride. During this time, participant will be asked about their pain and any side effects they may be having every 15 minutes for 2 hours and then every 30 minutes for another 2 hours. The study staff will also monitor participant's vital signs, and ask them a few more questions at the end of the study.

Length of Study Participation:

Although participant will stay in the emergency department for at least 4 hours, the average length of stay for participants with severe pain is about 9 hours. When participant is discharged from the emergency department or admitted to the hospital, their active participation in the study is over.

Follow-Up Phone Call:

About 24 hours after patient's active participation is over, the study nurse will call them to ask if they had any other side effects since taking part in the study. The phone call should last about 5 minutes. If participant is still an inpatient at the hospital, the study nurse may visit them and ask them these questions in person.

This is an investigational study. Hydromorphone hydrochloride is FDA approved and commercially available for the treatment of pain. Fentanyl nasal spray is FDA approved and commercially available for the treatment of pain. Its use to help with cancer pain in the emergency department is investigational.

Up to 84 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients with severe pain (i.e., >=7 on NRS, see Table 1) already on opioid therapy for one week or longer, at least 60 mg of oral morphine/day, 25 mcg of transdermal fentanyl/hour, 30 mg of oxycodone/day, 8 mg oral hydromorphone/day, 25 mg oral oxymorphone/day, or an equianalgesic dose of another opioid.
2. Ability to give informed consent before any trial-related activities (Trial-related activities are any procedure that would not have been performed during normal management of the subject.)
3. Ability and willingness to communicate the intensity of pain using NRS at the frequency dictated by the protocol

Exclusion Criteria:

1. Patients with a history of chronic active hepatitis, cirrhosis or hepatic encephalopathy
2. Inability to give informed consent
3. Known or suspected hypersensitivity or intolerance to fentanyl or hydromorphone or excipients in the study medications
4. Patients with sinusitis, obstruction of nasal passages, nasopharyngeal cancer, paranasal sinus malignancies, or any conditions in the nasopharyngeal anatomical area that may affect the absorption of fentanyl nasal spray.
5. Females who are pregnant, breast-feeding or intending to become pregnant. This exclusion criterion will be assessed by questioning the patient about the pregnancy status, breast-feeding status, the intent to become pregnant, the menopausal status, and the date of the last menstrual period.
6. Females of child-bearing potential, who are not using adequate contraceptive measures (including condoms, birth control pills, intrauterine devices, contraceptive implants, or other US FDA-approved contraceptives)
7. Previous participation in randomization in this trial
8. Has taken oral immediate release opioids within 4 hours prior to arrival.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-09-14 (Actual); Primary Completion 2020-06-21 (Actual); Study Completion 2020-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sai-Ching J. Yeung, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Banala SR, Khattab OK, Page VD, Warneke CL, Todd KH, Yeung SJ. Intranasal fentanyl spray versus intravenous opioids for the treatment of severe pain in patients with cancer in the emergency department setting: A randomized controlled trial. PLoS One. 2020 Jul 10;15(7):e0235461. doi: 10.1371/journal.pone.0235461. eCollection 2020. PMID 32649717
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cancer patients presenting to the M. D. Anderson Cancer Center Emergency Department for treatment of acute breakthrough pain, who met study inclusion criteria.
Pre-assignment Details: One (1) participant withdrew consent before treatment and 1 participant was found ineligible due to abnormal EKG.
Groups:
- Treatment Arm 1 (Intranasal Fentanyl): Fentanyl Nasal Spray 100mcg delivered at time 0 (defined as the time when intranasal Fentanyl spray is administered) with a rescue dose allowed at time 0.5 hour (h).
- Treatment Arm 2 (Intravenous Hydromorphone): Hydromorphone Hydrochloride 1.5mg pushed intravenously (IV) at time 0 (defined as the time of completion of opioid IV push) with a rescue dose allowed at time 0.5 hour (h).
- No Medication Administered: 1 Participant decided not to participate after signing the consent form; 1 Participant was found to have abnormal EKG changes with hypokalemia, hence removed from the study.
Period: Overall Study
Arm/Group | Treatment Arm 1 (Intranasal Fentanyl) | Treatment Arm 2 (Intravenous Hydromorphone) | No Medication Administered
Started | 42 | 40 | 2
Completed | 42 | 40 | 0
Not Completed | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Abnormal EKG changes | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm 1 (Intranasal Fentanyl) | Treatment Arm 2 (Intravenous Hydromorphone) | No Medication Administered | Total
Number analyzed (Participants) | 42 | 40 | 2 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 35 | 39 | 2 | 76
  >=65 years | 7 | 1 | 0 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.21 (14.452) | 50.33 (11.669) | 46 (1.000) | 52.32 (13.233)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 1 | 47
  Male | 19 | 17 | 1 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 6 | 0 | 17
  Not Hispanic or Latino | 31 | 34 | 2 | 67
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 3 | 1 | 14
  White | 31 | 35 | 1 | 67
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 40 | 2 | 84
Baseline NRS Pain Intensity [Mean (Standard Deviation); unit: NRS Pain Score] | 8.69 (1.093) | 8.95 (1.108) | NA (NA) — Data not collected | 8.82 (1.101)

OUTCOME MEASURES:

1. Primary Outcome: Non-inferiority of Fentanyl Nasal Spray Versus Intravenous Opioids in the Change in the Numeric Rating Scale (NRS) Pain Intensity Score at One Hour, Starting From the Time of Drug Delivery (Treatment Initiation).
Description: The median change in Numeric Rating Scale (NRS) pain intensity scores (assessed on an 11-point Likert scale with 0 = no pain and 10 = worst pain) from randomization, estimate of treatment initiation, to one hour post-treatment calculated for both treatment arms.
Time Frame: Baseline, One hour post time of drug delivery/treatment initiation
Measure: Median (Standard Deviation); unit: NRS Pain Intensity Score
Arm/Group | Treatment Arm 1 (Intranasal Fentanyl) | Treatment Arm 2 (Intravenous Hydromorphone)
Number analyzed (Participants) | 42 | 40
NRS Pain Intensity Score | 5.14 (2.16) | 4.90 (2.31)

2. Secondary Outcome: Number of Participants With Change in Numeric Rating Scale (NRS) Pain Intensity Score
Description: Change in NRS pain intensity scores from randomization to one hour after treatment start based on the percentage of participants with severe pain, NRS score = 7-10, one hour after treatment start for both treatment arms. Numeric Rating Scale (NRS) pain intensity scores (assessed on an 11-point Likert scale with 0 = no pain and 10 = worst pain).
Time Frame: One (1) hour after treatment start.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm 1 (Intranasal Fentanyl) | Treatment Arm 2 (Intravenous Hydromorphone)
Number analyzed (Participants) | 42 | 40
Participants | 5 | 10

ADVERSE EVENTS:
Time Frame: Within 24 hours after ED discharge or hospital admission
Description: No adverse events were reported prior to ED discharge or hospital admission.
Arm/Group | Treatment Arm 1 (Intranasal Fentanyl) | Treatment Arm 2 (Intravenous Hydromorphone) | No Medication Administered
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/40 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/40 | 0/2
Other Adverse Events (participants affected / at risk) | 1/42 | 3/40 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm 1 (Intranasal Fentanyl) (N=42) | Treatment Arm 2 (Intravenous Hydromorphone) (N=40) | No Medication Administered (N=2)
Headache (Nervous system disorders) | 1 | 3 | 0
Fatigue (General disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-21): https://cdn.clinicaltrials.gov/large-docs/64/NCT02459964/Prot_SAP_000.pdf